CLINICAL TRIAL: NCT06240208
Title: The Effects of Inactivity on GLP-1 Stimulated Appetite Regulation in Healthy Normal Weight Males: A Randomised, Parallel Group Study
Brief Title: Physical Inactivity and Appetite Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Grit Elster Legård, Primary Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-23055497
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inactivity (Experimental): Inactivity will be implemented as cessation of active commuting and all other structured exercise. Furthermore, steps will be reduced to a maximum of 1500 steps/day.
  Interventions: Behavioral: Inactivity
- Control (No Intervention): Participants will be instructed to maintain habitual physical activity and dietary habits.

INTERVENTIONS:
Behavioral: Inactivity — Inactivity will be implemented as cessation of active commuting and all other structured exercise. Furthermore, steps will be reduced to a maximum of 1500 steps/day.
  Arms: Inactivity

SUMMARY:
The goal of this parallel-group, two-arm, assessor-blinded, randomised clinical trial is to investigate the effects of reducing physical activity on food intake and satiety in physically active and healthy males, 40-55 years of age.

The main questions it aims to answer are:

* Does physical inactivity affect GLP-1 stimulated food intake?
* Does physical inactivity affect food preferences, satiety and other mechanisms supporting appetite regulation?

Participants will be randomised (1:1) to two weeks of either no intervention (control group) or inactivity. Inactivity will be implemented as cessation of active commuting and all other structured exercise. Furthermore, steps will be reduced to a maximum of 1500 steps/day.

Researchers will compare the inactivity group to the control group to see if physical inactivity impairs appetite regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age ≥ 40 years and ≤ 55 years
3. Body mass index (BMI) > 20 and < 25 kg/m2
4. Physical activity level should as a minimum include: Active commuting by biking a minimum of 10 km, four days per week or an equivalent amount of other physical activity four days per week.
5. Healthy (based on self-reporting, pre-study medical examination and biochemical screening)
6. Can adhere to two weeks of inactivity (refrain from running, cycling and all other exercise while reducing steps to max. 1500 pr. day)
7. Caucasian
8. No change in body weight > 5 kg within the last 6 months
9. Eats breakfast and lunch daily
10. Does not follow specific dietary restrictions
11. No disliking of spaghetti bolognese
12. No diagnosis of psychiatric disorder or treatment with anti-depressant or anti-psychotic medication
13. No history of suicidal behavior or ideations.
14. No previous surgical treatment for obesity
15. No cardiovascular disease
16. No rheumatologic disease
17. No metabolic/endocrine disease
18. No liver disease (ASAT or ALAT >2x upper normal range)
19. No other chronic disease
20. No elite sports
21. No frequent or chronic use of medications affecting bodyweight, physical performance, or inflammation (NSAIDS, DMARDS, corticosteroids)
22. No current infection
23. No history of cancer
24. No anemia (hematocrit <33%)
25. No smoking
26. No participation in other research intervention studies

Exclusion Criteria:

1. Clinical or biochemical signs of disease
2. HbA1c > 39 mmol/mol
3. Unable to allocate the needed time to fulfill the intervention
4. Language barrier, mental incapacity, unwillingness, or inability to understand and be able to complete the interventions

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The change in food intake at an ad libitum meal during GLP-1 infusion | From baseline (week 0) to follow-up (week 2).
  Food intake will be evaluated as ingested food in grams

SECONDARY OUTCOMES:
The change in preference for unhealthy food ( combined score for high fat food, savory food, and sweet food). | From baseline (week 0) to follow-up (week 2)
  Evaluated by visual food stimuli combined with eye tracking
The change in subjective experience of severity and type of food cravings | From baseline (week 0) to follow-up (week 2)
  Evaluated by the Control of Eating Questionnaire.
The change in subjective feeling of satiety | From baseline (week 0) to follow-up (week 2)
  Evaluated by a visual analogue scale
The change in subjective felling of hunger | From baseline (week 0) to follow-up (week 2)
  Evaluated by a visual analogue scale
The change in satiety composite appetite score | From baseline (week 0) to follow-up (week 2)
  Calculated from visual analog scales

OTHER OUTCOMES:
Change in secretion of gut hormones (GLP-1, GIP, PYY, ghrelin, CCK) | From baseline (week 0) to follow-up (week 2)
Change in gastric emptying rate | From baseline (week 0) to follow-up (week 2)
  Measured by surrogate marker paracetamol
Change in body composition (body weight, body mass index, lean mass, fat mass) | From baseline (week 0) to follow-up (week 2)
  Based on DXA scans
Change in physical fitness (maximal aerobic capacity, one repetition max) | From baseline (week 0) to follow-up (week 2)
Change in plasma glucose during ad libitum meal | From baseline (week 0) to follow-up (week 2)
  AUC (mol/hour)
Change in plasma insulin during ad libitum meal | From baseline (week 0) to follow-up (week 2)
  AUC (mol/h)
Change in plasma c-peptide during ad libitum meal | From baseline (week 0) to follow-up (week 2)
  AUC (mol/hour)
Change in glucagon supression during ad libitum meal | From baseline (week 0) to follow-up (week 2)
  The % glucagon supression at time 0-30min, 0-60min and 0-120min
Change in plasma insulin/glucagon ratio during ad libitum meal | From baseline (week 0) to follow-up (week 2)
  Insulin/glucagon at time=30, 60 and 120
Change in plasma glucose during mixed meal tolerance test | From baseline (week 0) to follow-up (week 2)
  AUC (mol/hour)
Change in plasma insulin during mixed meal tolerance test | From baseline (week 0) to follow-up (week 2)
  AUC (mol/hour)
Change in insulin/c-peptide ratio during mixed meal tolerance test | From baseline (week 0) to follow-up (week 2)
  Insulin/glucagon at time 30min, 60min, 120min and 180
Change in plasma c-peptide during mixed meal tolerance test | From baseline (week 0) to follow-up (week 2)
  AUC (mol/hour)
Change in glucagon supression during mixed meal tolerance test | From baseline (week 0) to follow-up (week 2)
  The % glucagon supression at time 0-30min, 0-60min, 0-120min and 0-180
Change in plasma insulin/glucagon ratio during mixed meal tolerance test | From baseline (week 0) to follow-up (week 2)
  Insulin/glucagon at time 30min, 60min, 120min and 180
Change in plasma concentration of cytokines (IL-1Ra, IL-6, IL-10, CRP, TNF-α, GDF-15) | From baseline (week 0) to follow-up (week 2)
Change in plasma concentration of adipokines (leptin and adiponectin) | From baseline (week 0) to follow-up (week 2)
Change in glycaemic variability | From baseline (week 0) to follow-up (week 2)
  CV% derived from free-living continuous glucose monitoring
Change in glycaemic variability | From baseline (week 0) to follow-up (week 2)
  SD derived from free-living continuous glucose monitoring
Change in glycaemic variability | From baseline (week 0) to follow-up (week 2)
  Mean glucose derived from free-living continuous glucose monitoring
Change in glycaemic variability | From baseline (week 0) to follow-up (week 2)
  Time in range derived from free-living continuous glucose monitoring
Change in physical and mental well-being | From baseline (week 0) to follow-up (week 2)
  Based on scores from WHO5, HAM-DS-S, and GAD-10 questionnaires
Change in physical and mental well-being | From baseline (week 0) to follow-up (week 2)
  Based on scores from WHO5 questionnaires
Change in symptoms of depression | From baseline (week 0) to follow-up (week 2)
  Based on scores from HAM-D6-S questionnaires
Change in symptoms of anxiety | From baseline (week 0) to follow-up (week 2)
  Based on scores from GAD-10 questionnaires
Change in sleep Quality | From baseline (week 0) to follow-up (week 2)
  Based on scores from Pittsburgh Sleep Quality Index
Change in plasma peptides | From baseline (week 0) to follow-up (week 2)
  Evaluated by peptidomics
Change in plasma metabolites | From baseline (week 0) to follow-up (week 2)
  Evaluated by metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Grit Elster Legård, MD, PhD, Principal Investigator — Centre for Physical Activity Research, Rigshospitalet
Locations (1):
- Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
If the data can be fully anonymized the data can be shared